CLINICAL TRIAL: NCT03493711
Title: Microbiota Differences Between Breastfed and Formula Fed Infants
Brief Title: Differences Between Breastfed and Formula Fed Infants
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 217562
Record Dates: First submitted 2018-02-12; First posted 2018-04-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, stool, breast milk, cheek swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast Fed: Exclusively breastfed for first 3 months of life
- Milk-based formula fed: Exclusively on Similac Advance Formula for at least 1 month prior to visit

SUMMARY:
This study will help us learn how a child's diet affects growth and development.

DETAILED DESCRIPTION:
This study will see how infants diet affects their growth and development. Up to 170 infants will be enrolled for one visit.

ELIGIBILITY:
Inclusion Criteria:

* Exclusive breast feeding or cow milk formula feeding during the first 3 months of life.
* For formula feeders, exclusively on Similac Advance Formula for at least 1 month prior to visit
* Age 2.5-3.5 months

Exclusion Criteria:

* Infants born to mother with preexisting medical conditions.
* Infants born to mother with medications during pregnancy known to influence fetal growth.
* Infants born to smoking, alcohol drinking or drug use mothers during pregnancy.
* Preterm

Ages: 2 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
The role of microbiota in gut | 2.5-3 months
  Stool samples will be collected
The role of microbiota in immune system development | 2.5-3 months
  Stool samples will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, RD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States